CLINICAL TRIAL: NCT03072537
Title: CrescNet - Computer-guided, Population-based Surveillance System for Growth Disorders
Brief Title: CrescNet - Growth Monitoring Network
Acronym: CrescNet
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Antje Koerner, Prof. Dr. med., Prof. Dr. med. Antje Körner, University of Leipzig
Other Study IDs: CrescNet
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Child Development; Growth Disorders
Keywords: growth; BMI; obesity; childhood; adolescence; development
MeSH Terms: conditions — Obesity; Growth Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CrescNet is a network of primary care physicians and pediatricians (n=219) and endocrinological treatment centers (n=33), established in Leipzig in 1998, whose aim is to improve the early detection of growth disorders. Secondary to this clinical aim, epidemiological analyses, for example on secular trends of growth data of children, are performed.

DETAILED DESCRIPTION:
Pediatricians participating in CrescNet provide pseudononymized data on patients' height, weight, and head circumferences to the CrescNet registry. Growth data are evaluated by automatized filter algorithms and by a pediatric endocrinologist. CrescNet does not have access to patients or personal patient data. Each participating pediatrician receives a quarterly screening report with recommendations for the work-up of children with abnormal growth or abnormal development of weight or body mass index.

The data registry is used for scientific purposes.The collection of data from healthy children allows the generation of evidence based statements about prevalence rates of growth disorders and also about the rates in disorders of weight development. For this, data are provided completely anonymized without allowing conclusions on personal patient data.

ELIGIBILITY:
Inclusion Criteria: Population based sample with inclusion of any patient seen by primary care or institutional physician/pediatrician, regardless of the objective for the visit (well child visits, acute visits or special requests)

Exclusion Criteria: none

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 479, 576 boys with 2,570, 041 visits und 453,510 girls with 2,427,350 visits from screening and/or consulting visits at 1 of the 435 participating German pediatricians.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 1998-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
growth disorders | 18 years
  Early detection of growth disorders in childhood and adolescent development. For this, not only absolute data but also growth velocity data are evaluated.
obesity | 18 years
  detection of critical age periods for the development of obesity. For this, not only absolute data but also growth velocity data are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Roland W Pfäffle, MD, Principal Investigator — University of Leipzig
Locations (1):
- CrescNet - University of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herget S, Markert J, Petroff D, Gausche R, Grimm A, Hilbert A, Kiess W, Bluher S. Psychosocial Well-Being of Adolescents Before and After a 1-Year Telephone-Based Adiposity Prevention Study for Families. J Adolesc Health. 2015 Sep;57(3):351-4. doi: 10.1016/j.jadohealth.2015.05.014. PMID 26299563
- [Background] Wagner IV, Paetzold C, Gausche R, Vogel M, Koerner A, Thiery J, Arsene CG, Henrion A, Guettler B, Keller E, Kiess W, Pfaeffle R, Kratzsch J. Clinical evidence-based cutoff limits for GH stimulation tests in children with a backup of results with reference to mass spectrometry. Eur J Endocrinol. 2014 Sep;171(3):389-97. doi: 10.1530/EJE-14-0165. Epub 2014 Jun 24. PMID 24966174
- [Background] Markert J, Alff F, Zschaler S, Gausche R, Kiess W, Bluher S. Prevention of childhood obesity: recruiting strategies via local paediatricians and study protocol for a telephone-based counselling programme. Obes Res Clin Pract. 2013 Dec;7(6):e476-86. doi: 10.1016/j.orcp.2012.07.008. PMID 24308890
- [Background] Alff F, Markert J, Zschaler S, Gausche R, Kiess W, Bluher S. Reasons for (non)participating in a telephone-based intervention program for families with overweight children. PLoS One. 2012;7(4):e34580. doi: 10.1371/journal.pone.0034580. Epub 2012 Apr 3. PMID 22509327
- [Background] Keller A, Klossek A, Gausche R, Hoepffner W, Kiess W, Keller E. [Selective primary obesity prevention in children]. Dtsch Med Wochenschr. 2009 Jan;134(1-2):13-8. doi: 10.1055/s-0028-1105883. Epub 2008 Dec 17. German. PMID 19090446
- [Background] Keller E, Gausche R, Meigen C, Keller A, Burmeister J, Kiess W. Auxological computer based network for early detection of disorders of growth and weight attainment. J Pediatr Endocrinol Metab. 2002 Feb;15(2):149-56. doi: 10.1515/jpem.2002.15.2.149. PMID 11874179
- [Background] Kiess W, Gausche R, Keller A, Burmeister J, Willgerodt H, Keller E. Computer-guided, population-based screening system for growth disorders (CrescNet) and on-line generation of normative data for growth and development. Horm Res. 2001;56 Suppl 1:59-66. doi: 10.1159/000048137. PMID 11786688
- [Background] Keller E, Burmeister J, Gausche R, Keller A, Hermanussen M, Kiess W. [Model program for the early detection and optimal treatment of disorders of growth and physical development using a medical competence netwok]. Z Arztl Fortbild Qualitatssich. 2000 Sep;94(8):695-8. German. PMID 11084726
- [Result] Kapellen TM, Gausche R, Dost A, Wiegand S, Flechtner-Mors M, Keller E, Kiess W, Holl RW; DPV-Science-Initiative of the German Competence Network Diabetes and the German Competence Network Obesity (Consortium LARGE). Children and adolescents with type 1 diabetes in Germany are more overweight than healthy controls: results comparing DPV database and CrescNet database. J Pediatr Endocrinol Metab. 2014 Mar;27(3-4):209-14. doi: 10.1515/jpem-2013-0381. PMID 24197766
- [Result] Miersch A, Vogel M, Gausche R, Siekmeyer W, Pfaffle R, Dittrich K, Kiess W. Blood pressure tracking in children and adolescents. Pediatr Nephrol. 2013 Dec;28(12):2351-9. doi: 10.1007/s00467-013-2596-3. PMID 23959541
- [Result] Hoepffner W, Pfaffle R, Gausche R, Meigen C, Keller E. Early detection of growth disorders with the CrescNet system at the Leipzig treatment center. Dtsch Arztebl Int. 2011 Feb;108(8):123-8. doi: 10.3238/arztebl.2011.0123. Epub 2011 Feb 25. PMID 21403802
- [Result] Bluher S, Meigen C, Gausche R, Keller E, Pfaffle R, Sabin M, Werther G, Odeh R, Kiess W. Age-specific stabilization in obesity prevalence in German children: a cross-sectional study from 1999 to 2008. Int J Pediatr Obes. 2011 Jun;6(2-2):e199-206. doi: 10.3109/17477166.2010.526305. Epub 2010 Nov 23. PMID 21091288
- [Result] Heger S, Korner A, Meigen C, Gausche R, Keller A, Keller E, Kiess W. Impact of weight status on the onset and parameters of puberty: analysis of three representative cohorts from central Europe. J Pediatr Endocrinol Metab. 2008 Sep;21(9):865-77. doi: 10.1515/JPEM.2008.21.9.865. PMID 18924580
- [Result] Meigen C, Keller A, Gausche R, Kromeyer-Hauschild K, Bluher S, Kiess W, Keller E. Secular trends in body mass index in German children and adolescents: a cross-sectional data analysis via CrescNet between 1999 and 2006. Metabolism. 2008 Jul;57(7):934-9. doi: 10.1016/j.metabol.2008.02.008. PMID 18555834
- [Result] Korner A, Kratzsch J, Gausche R, Schaab M, Erbs S, Kiess W. New predictors of the metabolic syndrome in children--role of adipocytokines. Pediatr Res. 2007 Jun;61(6):640-5. doi: 10.1203/01.pdr.0000262638.48304.ef. PMID 17426657
- [Result] Beger C, Merker A, Mumm R, Gausche R. Growth prediction of small for gestational age infants within the first weeks after birth. Anthropol Anz. 2018 Jun 11;74(5):377-382. doi: 10.1127/anthranz/2018/0820. Epub 2018 Feb 20. PMID 29461564
- [Result] Kess A, Spielau U, Beger C, Gausche R, Vogel M, Lipek T, Korner A, Pfaffle R, Kiess W. Further stabilization and even decrease in the prevalence rates of overweight and obesity in German children and adolescents from 2005 to 2015: a cross-sectional and trend analysis. Public Health Nutr. 2017 Dec;20(17):3075-3083. doi: 10.1017/S1368980017002257. Epub 2017 Sep 21. PMID 28931448
- [Result] Thiele AG, Gausche R, Lindenberg C, Beger C, Arelin M, Rohde C, Mutze U, Weigel JF, Mohnike K, Baerwald C, Scholz M, Kiess W, Pfaffle R, Beblo S. Growth and Final Height Among Children With Phenylketonuria. Pediatrics. 2017 Nov;140(5):e20170015. doi: 10.1542/peds.2017-0015. PMID 29089407
- [Derived] Vogel M, Geserick M, Gausche R, Beger C, Poulain T, Meigen C, Korner A, Keller E, Kiess W, Pfaffle R. Age- and weight group-specific weight gain patterns in children and adolescents during the 15 years before and during the COVID-19 pandemic. Int J Obes (Lond). 2022 Jan;46(1):144-152. doi: 10.1038/s41366-021-00968-2. Epub 2021 Sep 23. PMID 34556774
- [Derived] Geserick M, Vogel M, Gausche R, Lipek T, Spielau U, Keller E, Pfaffle R, Kiess W, Korner A. Acceleration of BMI in Early Childhood and Risk of Sustained Obesity. N Engl J Med. 2018 Oct 4;379(14):1303-1312. doi: 10.1056/NEJMoa1803527. PMID 30281992
- See also: Homepage CrescNet — http://crescnet.org/
- See also: Center for Pediatric Research Leipzig (CPL) — http://kik.uniklinikum-leipzig.de/kikcms.site,postext,arbeitsgruppen.html?PHPSESSID=4ka1kncm9nou..